CLINICAL TRIAL: NCT01324908
Title: T-regulatory Homing Subsets as a Predictor of Response in GVHD Treated With Extracorporeal Photopheresis
Brief Title: Biomarkers in Predicting Response in Patients With Graft-Versus-Host Disease Undergoing Extracorporeal Photophoresis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Byrne, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC CTT 1063; NCI-2011-00225 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-03-07; First posted 2011-03-29 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Graft Versus Host Disease (GVHD)
MeSH Terms: conditions — Graft vs Host Disease | interventions — Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Treg predictor of response to ECP) (Experimental): Patients undergo ECP twice a week for 4 weeks and then twice a week every 2 weeks for 8 weeks.
  Interventions: Procedure: extracorporeal photopheresis; Other: laboratory biomarker analysis

INTERVENTIONS:
Procedure: extracorporeal photopheresis — Undergo ECP
  Other Names: extracorporeal photophoresis
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies biomarkers in predicting response in patients with graft-versus-host disease (GVHD) undergoing extracorporeal photopheresis (ECP). ECP treats the patient's blood with ultraviolet light outside the body and kills the white blood cells before returning blood back into the patient's body. Studying samples of blood from patients with GVHD may help doctors identify and learn more about biomarkers related to GVHD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To show that extracorporeal photopheresis (ECP)increases skin and gut homing T regulatory (T-reg) cells in patients with GVHD clinically responding to ECP.

SECONDARY OBJECTIVES:

I. Response rates of GVHD with extracorporeal photopheresis(ECP)as measured by NIH response criteria

II. Incidence of T-reg cell frequency(%)with various NIH subtypes of chronic graft-versus-host disease (GVHD)

III. Incidence of T-reg homing subsets(%)with various NIH subtypes of chronic graft-versus-host disease (GVHD)

OUTLINE:

Patients undergo ECP twice a week for 4 weeks and then twice a week every 2 weeks for 8 weeks.

After completion of study treatment, patients are followed up at 2, 4, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any NIH subtype of chronic GVHD that is being treated with ECP
* Karnofsky Performance Scale (KPS) > 60% at time of study enrollment
* Life expectancy > 3 months
* Steroid dose not greater than 2 mg/kg prednisone equivalent at time of study enrollment
* If patient has steroid refractory GVHD (defined as worsening of GVHD after 3 days of 2 mg/kg prednisone equivalent or no improvement after 7 days of 2 mg/kg prednisone equivalent), time interval from start of steroids to initiation of ECP should not be > 14 days
* No use of an investigational agent within 2 weeks of starting ECP
* No uncontrolled bacterial, fungal or viral disease (therapy for cytomegalovirus [CMV] viremia is permitted)
* No evidence of relapse or progression of underlying disease (molecular evidence of relapse/progression or mixed chimerism is permitted)
* Women of childbearing potential (WOCBP) should be willing to use 2 forms of contraception; male patients should be willing to use contraception
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care

Exclusion Criteria:

* Female patients who are breastfeeding or pregnant
* Patients known to be human immunodeficiency virus (HIV) positive
* Bronchiolitis obliterans as the sole indication of ECP
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Mechanical ventilation, renal replacement therapy, admitted in intensive care until at time of enrollment
* Stage 4 gastrointestinal GVHD as per Seattle-Glucksberg criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-07; Primary Completion 2017-07-28 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Association of frequency of skin and gut homing Tregs (%) in patients with chronic GVHD with response to ECP. | 6 months after last patient is on study

SECONDARY OUTCOMES:
Response rates of GVHD with ECP as measured by NIH response criteria | at 6 months
Incidence of T-reg cell frequency (%) with various NIH subtypes of chronic GVHD | at 6 months
Incidence of T-reg homing subsets (%) with various NIH subtypes of chronic GVHD | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Madan Jagasia, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Virginia Commonwealth University, Massey Cancer Center, Richmond, Virginia

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/